CLINICAL TRIAL: NCT03205540
Title: Comparison Efficacy of Analgesic Techniques: Continuous Epidural Analgesia Versus Bilateral Single-shot Adductor Canal Blocks in Patients Undergoing Bilateral Total Knee Arthroplasty
Brief Title: Epidural Analgesia vs Adductor Canal Block in Bilateral TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwimon Tangwiwat, Assistant professor, Anesthesiology department, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Si 245/2017
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Osteo Arthritis Knee
Keywords: Continuous epidural analgesia; Bilateral single-shot adductor canal blocks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural analgesia (Experimental): Lumbar continuous epidural block
  Interventions: Procedure: Continuous epidural block
- Bilateral ACB (Experimental): Ultrasound-guided bilateral adductor canal blocks
  Interventions: Procedure: Bilateral single-shot bilateral adductor canal blocks

INTERVENTIONS:
Procedure: Continuous epidural block — Continuous epidural block at level L2-3 or L3-4 with 0.0625% bupivacaine + fentanyl 2 mcg/ml infusion epidurally 5 ml/hr for 48 hours postoperatively.
  Arms: Epidural analgesia
Procedure: Bilateral single-shot bilateral adductor canal blocks — Bilateral single-shot adductor canal blocks, ultrasound guidance, with 0.33% bupivacaine 15 ml on each side.
  Arms: Bilateral ACB

SUMMARY:
This study evaluates postoperative analgesic efficacy within 48 hours between epidural analgesia and single-shot bilateral adductor canal blocks in bilateral total knee arthroplasty. Half of participants will be received continuous epidural analgesia, while other half of participants will be received single-shot bilateral adductor canal blocks.

DETAILED DESCRIPTION:
Continuous epidural analgesia is effective postoperative pain control but it has some limitations in patients with hypotension, concurrent anticoagulants, technical difficulty, urinary retention.

Adductor canal block is less invasive than continuous epidural analgesia. It provides effective analgesia for total knee arthroplasty and preserves quadriceps muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old undergoing bilateral total knee arthroplasty
* American Society of Anesthesiologists physical status classification 1-3

Exclusion Criteria:

* Participants deny to enroll the study
* Allergy to bupivacaine
* Weight less than 50 kilograms
* Hepatic disease
* Contraincation for neuraxial block or adductor canal block
* Uncontrolled cardiovascular disease
* Creatinine clearance less than 50 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
pain scores at rests | 48 hours postoperatively
  numerical rating scales

SECONDARY OUTCOMES:
morphine consumptions | 48 hours postoperatively
  total miligrams of morphine use in each arm
pain scores on movement | 48 hours postoperatively
  numerical rating scales
side effects of interventions | 48 hours postoperatively
  nausea vomiting hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Background] Dimitris CN, Taylor BC, Mowbray JG, Steensen RN, Gaines ST. Perioperative morbidity and mortality of 2-team simultaneous bilateral total knee arthroplasty. Orthopedics. 2011 Dec 6;34(12):e841-6. doi: 10.3928/01477447-20111021-02. PMID 22146199
- [Background] Choi PT, Bhandari M, Scott J, Douketis J. Epidural analgesia for pain relief following hip or knee replacement. Cochrane Database Syst Rev. 2003;2003(3):CD003071. doi: 10.1002/14651858.CD003071. PMID 12917945
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Gerrard AD, Brooks B, Asaad P, Hajibandeh S, Hajibandeh S. Meta-analysis of epidural analgesia versus peripheral nerve blockade after total knee joint replacement. Eur J Orthop Surg Traumatol. 2017 Jan;27(1):61-72. doi: 10.1007/s00590-016-1846-z. Epub 2016 Sep 3. PMID 27592218
- [Background] Fowler SJ, Symons J, Sabato S, Myles PS. Epidural analgesia compared with peripheral nerve blockade after major knee surgery: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2008 Feb;100(2):154-64. doi: 10.1093/bja/aem373. PMID 18211990